CLINICAL TRIAL: NCT01289093
Title: Quality of Life After Laparoscopic Inguinal- Incisional- and Umbilical Herniotomy.
Brief Title: Quality of Life After Laparoscopic Inguinal- Incisional and Umbilical Herniotomy.
Acronym: life-in
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Bispebjerg Hospital (Other); University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Mette M W Christoffersen, MD, Zealand University Hospital
Other Study IDs: 1234
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Inguinal Hernia; Incisional Hernia; Umbilical Hernias
Keywords: inguinal hernia; incisional hernia; quality of life; disease-specific
MeSH Terms: conditions — Hernia, Inguinal; Incisional Hernia; Hernia, Umbilical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- laparoscopic ingunal herniotomy
- laparoscopic incisional herniotomy
- Lichtenstein inguinal herniotomy
- laparoscopic umbilical hernia repair

SUMMARY:
LIFE-IN. Quality of life after operation for hernias are not well investigated and lack a good and easy-to-understand-tool to measure it. Carolina Comfort Scale (CCS) is a disease-specific quality of life questionnaire, designed by an American group, to monitor quality of life in patients undergoing operation for hernias.

The investigators wish to test this questionnaire against Visual Analogue Scale (VAS) scores for core-hernia symptoms, to see if the CCS is a good way to monitor the changes in quality of life and other well-known core-symptoms before and after herniotomies.

DETAILED DESCRIPTION:
The investigators include consecutively all in all 140 patients. 100 with inguinal hernias; 50 who is getting a Lichtenstein operation and 50 who is getting a laparoscopic operation. Furthermore minimum 20 patients who is getting a laparoscopic operation for incisional hernia and minimum 20 who went through umbilical herniotomy. The investigators monitor their pain, sensation of mesh, movement limitations, over-all well-being, fatigue and life-quality, with both CCS and VAS questionnaires 5 times. One time preoperative and 4 times after operation, on the 1sth, 7th, 30th and 90th day after operation.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic and open operations for inguinal hernia
* elective laparoscopic operation for incisional- and umbilical hernia
* primary hernia
* uni-bilateral hernias and one or more incisional hernias

Exclusion Criteria:

* expected bad compliance to the study
* acute operations
* re-operations
* secondary operations
* primary operation with reoperation within 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
quality of life | before operation until 90 days postoperative
  pain, sensation of mesh, movement limitations, over-all well-being, fatigue and quality of life. These core symptoms will be measured 5 times with the 2 questionnaires CCS and VAS. One time before and 4 times after the operation with both the CCS and VAS, to see if the is a graphical correlation between the to questionnaires and to find out which of the two questionnaires is best.

SECONDARY OUTCOMES:
acceptability | preoperative untill 90 days postoperative
  The investigators measure the patients satisfaction with the instruments and which one (VAS or CCS) they prefer.

CONTACTS AND LOCATIONS:
Overall Officials: Thue Bisgaard, MD, Study Director — Zealand University Hospital
Locations (1):
- Koege University Hospital, Koege, Denmark